CLINICAL TRIAL: NCT06366087
Title: A Two-Period, Two-Sequence, Two-Treatment, Single-Dose Crossover Study of Atropine Sulfate Ophthalmic Solution (1%) Administered Sublingually vs Atropine Sulfate Administered Intramuscularly for Bioequivalence Determination
Brief Title: Sublingual Atropine Bioequivalence by Route of Administration (SABER)
Acronym: SABER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Collaborators: Rho Federal Systems Division, Inc. (Industry); Allucent Government Services (US), LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BP-C-24-001
Record Dates: First submitted 2024-04-11; First posted 2024-04-15 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Atropine Bioequivalence
Keywords: Pharmaceutical Solutions; Adjuvants, Anesthesia; Anti-Arrhythmia Agents; Bronchodilator Agents; Autonomic Agents; Peripheral Nervous System Agents; Physiological Effects of Drugs; Anti-Asthmatic Agents; Respiratory System Agents; Mydriatics; Parasympatholytics; Muscarinic Antagonists; Cholinergic Antagonists; Cholinergic Agents; Neurotransmitter Agents; Molecular Mechanisms of Pharmacological Action; Atropine; Ophthalmic Solutions
MeSH Terms: interventions — Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sublingual (Experimental): 1 mg (100 µL of a 1% w/v solution), administered SL by pipette with at least a 30 second dwell time without swallowing.
  Interventions: Drug: Atropine Sulfate Ophthalmic Solution USP, 1%
- Intramuscular (Active Comparator): Multidose vial presentation, 1 mg (2.5 ml) administered by IM injection into the mid-anterolateral thigh.
  Interventions: Drug: Atropine Sulfate Injection, USP 8 mg/20 mL (0.4 mg/mL)

INTERVENTIONS:
Drug: Atropine Sulfate Ophthalmic Solution USP, 1% — Atropine Sulfate Ophthalmic Solution, USP 1% manufactured by Bausch & Lomb Americas Inc., is a sterile topical anti-muscarinic indicated for mydriasis, cycloplegia, and penalization of the healthy eye to treat amblyopia. Each mL of Atropine Sulfate Ophthalmic Solution USP, 1% contains the active ingredient atropine sulfate 10 mg, equivalent to 8.3 mg of atropine. Inactive ingredients are boric acid, hydroxypropyl methylcellulose, and water for injection, USP; hydrochloric acid and/or sodium hydroxide may be added to adjust pH (3.5 to 6.0). Atropine Sulfate Ophthalmic Solution, USP 1% will be supplied in 0.4 mL single-dose vials and will be administered as a single dose to a single participant. 100 μL of Atropine Sulfate Ophthalmic Solution, USP 1% will be given sublingually by pipette to deliver 1.0 mg of atropine sulfate. Before administration, participants will be told to swallow. Once given, participants will be told to try not to swallow for 30 seconds and then swallow normally.
  Arms: Sublingual
Drug: Atropine Sulfate Injection, USP 8 mg/20 mL (0.4 mg/mL) — Atropine sulfate injection, USP is a muscarinic antagonist used for temporary blockade of severe/life-threatening muscarinic effects and to treat symptomatic bradycardia. Atropine Sulfate Injection, USP, 8 mg/20 mL (0.4 mg/mL) manufactured by Fresenius Kabi is a sterile, nonpyrogenic, isotonic, clear solution of atropine sulfate in water for injection with sodium chloride sufficient to render the solution isotonic. Each mL contains atropine sulfate, 0.4 mg; benzyl alcohol, 9 mg; and sodium chloride 9 mg; it may also contain sulfuric acid for pH adjustment, pH 3.5 (3.0 to 3.8). Atropine Sulfate Injection, USP will be supplied in 8 mg/20 mL multidose vials (0.4 mg/mL). Each vial will be used to administer multiple doses to multiple participants. 2.5 mL will be injected into the mid-anterolateral thigh to deliver 1.0 mg of atropine sulfate. Vials will be dated/timed and will not be given after 24 hours of first entry.
  Arms: Intramuscular

SUMMARY:
A randomized, two-period, two-sequence, crossover study to assess the bioequivalence, bioavailability, and pharmacokinetics (PK) of a single dose of atropine administered sublingually (SL) or intramuscularly (IM) in healthy adult volunteers.

DETAILED DESCRIPTION:
This is a randomized, two-period, two-sequence, crossover study to assess the bioequivalence, bioavailability, and pharmacokinetics (PK) of a single dose of atropine administered SL or IM in healthy adult volunteers. A total of 46 healthy male and non-pregnant female volunteers will be randomized, with the goal of obtaining at least 36 evaluable participants in the per protocol population. Additional participants may be randomized if participants are withdrawn prior to receiving one or both doses of study drug. Eligible participants will be randomized at a 1:1 ratio to receive one of two treatment dosing sequences (A [Visit 1 SL, Visit 2 IM] or B [Visit 1 IM, Visit 2 SL]).

Volunteers will be screened for study participation from Days -14 to -3. Eligible participants will be enrolled and randomized to receive one of two dosing sequences (Sequence A or Sequence B) until the target enrollment for the study is met. Once randomized, each participant will receive 2 doses of atropine separated by a wash out period of 6 ±1 days. During Visit 1 (Day 1) and Visit 2 (Day 8), participants will be administered SL or IM atropine, according to their randomly assigned dosing sequence. At each dosing visit, blood samples for PK will be collected at time 0 (pre-dose) and at 13 time points post-dose at 5, 10, 15, 20, 30, 45, 60, and 90 minutes and 2, 2.5, 4, 6, and 8 hours after dosing. Participants will be discharged from the clinic after the 8-hour blood sample collection. Participants will be followed for approximately 6 days after their last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and non-pregnant female volunteers between the ages of 18 and 65 years, inclusive, at time of consent.
2. Willing and able to provide written informed consent.
3. Females who are of childbearing potential and are sexually active with a male partner must have used an adequate method of birth control for at least 2 months prior to Screening and must agree to continue using an adequate method of birth control from Screening through Follow-up (Day 15).

   1. A female of childbearing potential is defined as a post onset of menarche and premenopausal female capable of becoming pregnant. This does not include females who meet any of the following conditions: menopausal >2 years, tubal ligation >1 year, bilateral salpingo-oophorectomy, or hysterectomy.
   2. Adequate contraception is defined as a contraceptive method with a failure rate of less than 1% per year when used consistently and correctly and when applicable, in accordance with the product label. Examples include oral contraceptives, injectable progestogen, implants of etonogestrel or levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, intrauterine device or intrauterine system, or male partner sterilization at least 6 months prior to the participant's Screening Visit.
4. In the judgment of the investigator, the participant is in good health, based on review of medical history and the results of Screening evaluation (including vital signs, physical examination, 12-lead electrocardiogram [ECG], and Screening laboratory assessments, performed no more than 14 days prior to randomization into the study).
5. Able to comply with the dosing instructions and available to complete the study Schedule of Assessments.

Exclusion Criteria:

1. Females who have a positive pregnancy test or who are breastfeeding.
2. Participants with thyroid disease as evidenced by a thyroid-stimulating hormone (TSH) <0.9 × lower limit of normal (LLN) or > 1.2 × upper limit of normal (ULN) at Screening (This Screening test will not be repeated prior to subsequent dosing).
3. Participants with aspartate aminotransferase (AST), alanine aminotransferase (ALT), or serum creatinine >1.5 × ULN at Screening. (These Screening tests will not be repeated prior to subsequent dosing.)
4. Have known human immunodeficiency virus (HIV), or acute or chronic hepatitis B or hepatitis C infection based on medical history; or test positive for any of these at Screening. Participants who have been effectively treated for hepatitis C, as evidenced by a negative hepatitis C RNA confirmation test and who no longer require antiviral therapy, are eligible for participation. (These Screening tests will not be repeated prior to subsequent dosing.)
5. Participants who took any prescription medications (with the exception of oral contraceptives or hormone replacement therapy) within 30 days of Screening. Prior to each dose, the investigator will review prohibited medication use and determine whether the participant should be terminated from further dosing.
6. Participants who took any over-the-counter medication/vitamins/herbal supplements in the last 72 hours prior to Screening. Prior to each dose, the investigator will review prohibited medication use and determine whether the participant should be terminated from further dosing.
7. Participants who are current smokers or are currently using any oral nicotine/oral tobacco product (e.g. snuff, chew, lozenges, nicotine gum, pouches) or electronic cigarette or vaping device (e.g., e-cigarette, mod, vape pen, JUUL, e-cigar, e-hookah, e-pipe, vape pods) or have used any of these products within 6 months prior to Screening.
8. Participants with glaucoma and/or history of ocular surgery (including LasikTM), ocular trauma, or congenital ocular disorder.
9. Participants with any history of heart disease, including but not limited to hypertension, coronary artery disease, arrhythmia (treated or untreated), congestive heart failure, pacemaker, history of vasovagal syncope, any supraventricular tachycardia, peripheral vascular disease, or claudication.
10. Participants with clinically significant arrhythmias or abnormal conduction; abnormal conduction is defined as a prolonged PR or QRS, or a QTc ≥450 msec for males or ≥470 msec for females.
11. Participants with a history of partial organic pyloric stenosis, chronic constipation, gastroparesis, or other gastrointestinal motility issues.
12. Participants with a history of xerostomia due to an underlying disease or previous radiation therapy to the head and neck.
13. Males with history of symptomatic prostatic hypertrophy; males or females with a history of urinary hesitancy or retention.
14. Participants with a blood pressure >140/90 mm Hg taken after the participant has been seated and resting for at least five minutes.
15. Participants with a history or current diagnosis of myasthenia gravis.
16. Participants who have donated blood within 8 weeks of Screening or intend to donate blood during the study period.
17. Participants with a history of drug or alcohol abuse in the last two years or evidence of a positive urine drug test at Screening. (This Screening test will not be repeated prior to subsequent dosing.)
18. Participants with a known sensitivity or prior adverse reaction to atropine.
19. Participants who have consumed alcohol within 24 hours prior to each Pre-dose Visit. (This will be assessed only at Visit 1 [Pre-dose] and Visit 2 [Pre-dose].)
20. Participants with any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled, would interfere with SL or IM administration of study drug, or would otherwise interfere with interpretation of study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Eisnor, MD, Study Chair — Biomedical Advanced Research and Development Authority; Michael Schwartz, MD, Study Chair — Biomedical Advanced Research and Development Authority
Locations (1):
- Johnson County Clin-Trials (JCCT), Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single US site between April 2024 and May 2024. Potential participants signed informed consent before undergoing any screening procedures to confirm eligibility.
Pre-assignment Details: Of 107 consented participants, 46 eligible participants were enrolled and randomized to treatment. Of the remaining 61 consented participants, 40 participants did not meet eligibility criteria, and 21 participants were not enrolled or randomized due to enrollment/randomization targets having already been met.
Groups:
- Sequence A: Atropine Sulfate Sublingual - Atropine Sulfate Intramuscular: Participants dosed sublingually (SL) on Visit 1 (Day 1) and dosed intramuscularly (IM) on Visit 2 (Day 8).
- Sequence B: Atropine Sulfate Intramuscular - Atropine Sulfate Sublingual: Participants dosed intramuscularly (IM) on Visit 1 (Day 1) and dosed sublingually (SL) on Visit 2 (Day 8).
Period: Overall Study
Arm/Group | Sequence A: Atropine Sulfate Sublingual - Atropine Sulfate Intramuscular | Sequence B: Atropine Sulfate Intramuscular - Atropine Sulfate Sublingual
Started | 23 | 23
Completed | 23 | 22
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A: Atropine Sulfate Sublingual - Atropine Sulfate Intramuscular | Sequence B: Atropine Sulfate Intramuscular - Atropine Sulfate Sublingual | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (11.64) | 41.4 (14.65) | 41.9 (13.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 14 | 9 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 20 | 21 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 10 | 7 | 17
  White | 10 | 11 | 21
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: The Bioequivalence of Atropine Sulfate Administered SL Versus Administered IM as Measured by Area Under the Analyte Concentration Versus Time Curve to Infinity (AUCinf).
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 5, 10, 15, 20, 30, 45, 60, and 90 minutes, and 2, 2.5, 4, 6, and 8 hours. PK parameters were estimated for each subject and route using noncompartmental analysis (NCA) methods. AUCinf is summarized by route of administration as the geometric mean and coefficient of variation of the geometric mean for all evaluable participants and expressed as min*ng/mL. Geometric ratios of least-square means and associated 90% confidence intervals are reported from a linear mixed model. Bioequivalence will be considered met if the 90% CI of the ratio for AUCinf lies within 80.00 to 125.00%.
Time Frame: Pre-dose through 8 hours post-dose at Days 1 and 8
Population: PK Analysis Population includes all participants who are randomized, receive at least 1 study drug dose, and have PK samples collected for that period. Participants needed to have plasma concentration results at 3 or more time points beyond tmax (time to maximum measured plasma concentration) in order to have an evaluable estimate for AUCinf.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*ng/mL
Groups:
- Sublingual: Atropine Sulfate Ophthalmic Solution, USP 1% manufactured by Bausch & Lomb Americas Inc., is a sterile topical anti-muscarinic indicated for mydriasis, cycloplegia, and penalization of the healthy eye to treat amblyopia. Each mL of Atropine Sulfate Ophthalmic Solution USP, 1% contains the active ingredient atropine sulfate 10 mg, equivalent to 8.3 mg of atropine. Inactive ingredients are boric acid, hydroxypropyl methylcellulose, and water for injection, USP; hydrochloric acid and/or sodium hydroxide may be added to adjust pH (3.5 to 6.0). Atropine Sulfate Ophthalmic Solution, USP 1% will be supplied in 0.4 mL single-dose vials and will be administered as a single dose to a single participant. 100 μL of Atropine Sulfate Ophthalmic Solution, USP 1% will be given sublingually by pipette to deliver 1.0 mg of atropine sulfate. Before administration, participants will be told to swallow. Once given, participants will be told to try not to swallow for 30 seconds and then swallow normally.
- Intramuscular: Atropine sulfate injection, USP is a muscarinic antagonist used for temporary blockade of severe/life-threatening muscarinic effects and to treat symptomatic bradycardia. Atropine Sulfate Injection, USP, 8 mg/20 mL (0.4 mg/mL) manufactured by Fresenius Kabi is a sterile, nonpyrogenic, isotonic, clear solution of atropine sulfate in water for injection with sodium chloride sufficient to render the solution isotonic. Each mL contains atropine sulfate, 0.4 mg; benzyl alcohol, 9 mg; and sodium chloride 9 mg; it may also contain sulfuric acid for pH adjustment, pH 3.5 (3.0 to 3.8). Atropine Sulfate Injection, USP will be supplied in 8 mg/20 mL multidose vials (0.4 mg/mL). Each vial will be used to administer multiple doses to multiple participants. 2.5 mL will be injected into the mid-anterolateral thigh to deliver 1.0 mg of atropine sulfate. Vials will be dated/timed and will not be given after 24 hours of first entry.
Arm/Group | Sublingual | Intramuscular
Number analyzed (Participants) | 41 | 46
min*ng/mL | 562.456 (23.0) | 814.860 (19.0)
Statistical Analysis 1: Comparison: Sublingual vs Intramuscular; Test type: Other — Estimation only. Estimates are back-transformed and based on a random effects linear model with log10 numeric response variable, adjusting for study route received, dosing sequence, and period, with a random effect for subject nested within dosing sequence; Mixed Models Analysis; Ratio of geometric least-square means = 0.70, 90% CI 2-sided [0.670 to 0.724] — Bioequivalence will be considered met if the 90% CI of the ratio for AUCinf lies within 80.00 to 125.00%

2. Primary Outcome: The Bioequivalence of Atropine Sulfate Administered SL Versus Administered IM as Measured by Area Under the Analyte Concentration Versus Time Curve to Time of Last Quantifiable Data Point (AUCt).
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 5, 10, 15, 20, 30, 45, 60, and 90 minutes, and 2, 2.5, 4, 6, and 8 hours. PK parameters were estimated for each subject and route using noncompartmental analysis (NCA) methods. AUCt is summarized by route of administration as the geometric mean and coefficient of variation of the geometric mean for all evaluable participants and expressed as min*ng/mL. Geometric ratios of least-square means and associated 90% confidence intervals are reported from a linear mixed model. Bioequivalence will be considered met if the 90% CI of the ratio for AUCt lies within 80.00 to 125.00%.
Time Frame: Pre-dose through 8 hours post-dose at Days 1 and 8
Population: PK Analysis Population includes all participants who are randomized, receive at least 1 study drug dose, and have PK samples collected for that period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*ng/mL
Arm/Group | Sublingual | Intramuscular
Number analyzed (Participants) | 45 | 46
min*ng/mL | 456.944 (22.7) | 683.672 (20.5)
Statistical Analysis 1: Comparison: Sublingual vs Intramuscular; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of geometric least-square means = 0.67, 90% CI 2-sided [0.640 to 0.697] — Bioequivalence will be considered met if the 90% CI of the ratio for AUCt lies within 80.00 to 125.00%

3. Secondary Outcome: AUC45 - The Relative Bioavailability (Plasma Concentrations) of Atropine Sulfate Administered SL Versus IM as Measured by Area Under the Analyte Concentration Versus Time Curve to Time 45 Minutes (AUC45)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 5, 10, 15, 20, 30, 45, 60, and 90 minutes, and 2, 2.5, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using noncompartmental analysis (NCA) methods.
  AUC45 is summarized by route of administration as the geometric mean and coefficient of variation for the geometric mean for all evaluable participants expressed as min*ng/mL. Geometric ratios of least-square means and associated 90% confidence intervals are reported from a linear mixed model
Time Frame: 0 hour (pre-dose), 5, 10, 15, 20, 30, and 45 minutes post-dose on Days 1 and 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*ng/mL
Arm/Group | Sublingual | Intramuscular
Number analyzed (Participants) | 45 | 46
min*ng/mL | 11.559 (98.9) | 106.046 (34.9)
Statistical Analysis 1: Comparison: Sublingual vs Intramuscular; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of geometric least-square means = 0.11, 90% CI 2-sided [0.088 to 0.136]

4. Secondary Outcome: AUC60 - The Relative Bioavailability (Plasma Concentrations) of Atropine Sulfate Administered SL Versus IM as Measured by Area Under the Analyte Concentration Versus Time Curve to Time 60 Minutes (AUC60)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 5, 10, 15, 20, 30, 45, 60, and 90 minutes, and 2, 2.5, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using noncompartmental analysis (NCA) methods.
  AUC60 is summarized by route of administration as the geometric mean and coefficient of variation for the geometric mean for all evaluable participants expressed as min*ng/mL. Geometric ratios of least-square means and associated 90% confidence intervals are reported from a linear mixed model.
Time Frame: 0 hour (pre-dose), 5, 10, 15, 20, 30, 45, and 60 minutes post-dose at Days 1 and 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*ng/mL
Arm/Group | Sublingual | Intramuscular
Number analyzed (Participants) | 45 | 46
min*ng/mL | 21.903 (103.1) | 145.215 (31.8)
Statistical Analysis 1: Comparison: Sublingual vs Intramuscular; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of geometric least-square means = 0.15, 90% CI 2-sided [0.120 to 0.189]

5. Secondary Outcome: AUC90 - The Relative Bioavailability (Plasma Concentrations) of Atropine Sulfate Administered SL Versus IM as Measured by Area Under the Analyte Concentration Versus Time Curve to Time 90 (AUC90)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 5, 10, 15, 20, 30, 45, 60, and 90 minutes, and 2, 2.5, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using noncompartmental analysis (NCA) methods.
  AUC90 is summarized by route of administration as the geometric mean and coefficient of variation for the geometric mean for all evaluable participants expressed as min*ng/mL. Geometric ratios of least-square means and associated 90% confidence intervals are reported from a linear mixed model.
Time Frame: 0 (pre-dose), 5, 10, 15, 20, 30, 45, 60, and 90 minutes post-dose at Days 1 and 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*ng/mL
Arm/Group | Sublingual | Intramuscular
Number analyzed (Participants) | 45 | 46
min*ng/mL | 56.521 (74.2) | 217.844 (27.8)
Statistical Analysis 1: Comparison: Sublingual vs Intramuscular; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of geometric least-square means = 0.26, 90% CI 2-sided [0.217 to 0.309]

6. Secondary Outcome: AUC120 - The Relative Bioavailability (Plasma Concentrations) of Atropine Sulfate Administered SL Versus IM as Measured by Area Under the Analyte Concentration Versus Time Curve to Time 120 Minutes (AUC120)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 5, 10, 15, 20, 30, 45, 60, and 90 minutes, and 2, 2.5, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using noncompartmental analysis (NCA) methods.
  AUC120 is summarized by route of administration as the geometric mean and coefficient of variation for the geometric mean for all evaluable participants expressed as min*ng/mL. Geometric ratios of least-square means and associated 90% confidence intervals are reported from a linear mixed model.
Time Frame: 0 (pre-dose), 5, 10, 15, 20, 30, 45, 60, 90, and 120 minutes post-dose at Days 1 and 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*ng/mL
Arm/Group | Sublingual | Intramuscular
Number analyzed (Participants) | 45 | 46
min*ng/mL | 103.146 (52.9) | 283.847 (25.8)
Statistical Analysis 1: Comparison: Sublingual vs Intramuscular; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of geometric least-square means = 0.36, 90% CI 2-sided [0.318 to 0.416]

7. Secondary Outcome: AUC150 - The Relative Bioavailability (Plasma Concentrations) of Atropine Sulfate Administered SL Versus IM as Measured by Area Under the Analyte Concentration Versus Time Curve to Time 150 Minutes (AUC150)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 5, 10, 15, 20, 30, 45, 60, and 90 minutes, and 2, 2.5, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using noncompartmental analysis (NCA) methods.
  AUC150 is summarized by route of administration as the geometric mean and coefficient of variation for the geometric mean for all evaluable participants expressed as min*ng/mL. Geometric ratios of least-square means and associated 90% confidence intervals are reported from a linear mixed model.
Time Frame: 0 (pre-dose), 5, 10, 15, 20, 30, 45, 60, 90, 120, and 150 minutes post-dose at Days 1 and 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*ng/mL
Arm/Group | Sublingual | Intramuscular
Number analyzed (Participants) | 45 | 46
min*ng/mL | 151.441 (41.5) | 343.066 (24.6)
Statistical Analysis 1: Comparison: Sublingual vs Intramuscular; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of geometric least-square means = 0.44, 90% CI 2-sided [0.396 to 0.492]

8. Secondary Outcome: AUC240 - The Relative Bioavailability (Plasma Concentrations) of Atropine Sulfate Administered SL Versus IM as Measured by Area Under the Analyte Concentration Versus Time Curve to Time 240 Minutes (AUC240)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 5, 10, 15, 20, 30, 45, 60, and 90 minutes, and 2, 2.5, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using noncompartmental analysis (NCA) methods.
  AUC240 is summarized by route of administration as the geometric mean and coefficient of variation for the geometric mean for all evaluable participants expressed as min*ng/mL. Geometric ratios of least-square means and associated 90% confidence intervals are reported from a linear mixed model.
Time Frame: 0 (pre-dose), 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, and 240 minutes post-dose at Days 1 and 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*ng/mL
Arm/Group | Sublingual | Intramuscular
Number analyzed (Participants) | 45 | 46
min*ng/mL | 275.948 (27.5) | 484.704 (22.7)
Statistical Analysis 1: Comparison: Sublingual; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of geometric least-square means = 0.57, 90% CI 2-sided [0.532 to 0.608]

9. Secondary Outcome: The Relative Bioavailability of Atropine Sulfate Administered SL Versus IM as Measured by Maximum Measured Plasma Concentration (Cmax)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 5, 10, 15, 20, 30, 45, 60, and 90 minutes, and 2, 2.5, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using noncompartmental analysis (NCA) methods.
  Cmax is summarized by route of administration as the geometric mean and coefficient of variation of the geometric mean for all evaluable participants and expressed as ng/mL. Geometric ratios of least-square means and associated 90% confidence intervals are reported from a linear mixed model.
Time Frame: Pre-dose through 8 hours post-dose at Days 1 and 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Sublingual | Intramuscular
Number analyzed (Participants) | 45 | 46
ng/mL | 1.805 (26.6) | 3.176 (35.0)
Statistical Analysis 1: Comparison: Sublingual vs Intramuscular; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of geometric least-square means = 0.57, 90% CI 2-sided [0.524 to 0.620]

10. Secondary Outcome: The Relative Bioavailability of Atropine Sulfate Administered SL Versus IM as Measured by Time to Cmax (Tmax)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 5, 10, 15, 20, 30, 45, 60, and 90 minutes, and 2, 2.5, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using noncompartmental analysis (NCA) methods.
  tmax is summarized by route of administration as the mean and standard deviation for all evaluable participants and expressed as minutes.
Time Frame: Pre-dose through 8 hours post-dose at Days 1 and 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Sublingual | Intramuscular
Number analyzed (Participants) | 45 | 46
min | 118.0 (49.19) | 34.3 (22.20)

11. Secondary Outcome: The Relative Bioavailability of Atropine Sulfate Administered SL Versus IM as Measured by Apparent Terminal Elimination Half-life (t1/2)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 5, 10, 15, 20, 30, 45, 60, and 90 minutes, and 2, 2.5, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using noncompartmental analysis (NCA) methods.
  t1/2 is summarized by route of administration as the mean and standard deviation for all evaluable participants and expressed as minutes.
Time Frame: Pre-dose through 8 hours post-dose at Days 1 and 8
Population: PK Analysis Population includes all participants who are randomized, receive at least 1 study drug dose, and have PK samples collected for that period. Participants needed to have plasma concentration results at 3 or more time points beyond tmax (time to maximum measured plasma concentration) in order to have an evaluable estimate for t1/2.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Sublingual | Intramuscular
Number analyzed (Participants) | 41 | 46
min | 171.089 (31.7096) | 175.682 (35.6344)

12. Secondary Outcome: The Relative Bioavailability of Atropine Sulfate Administered SL Versus IM as Measured by Terminal Elimination Rate Constant (λz)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 5, 10, 15, 20, 30, 45, 60, and 90 minutes, and 2, 2.5, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using noncompartmental analysis (NCA) methods.
  λz is summarized by route of administration as the mean and standard deviation for all evaluable participants and expressed as 1/min.
Time Frame: Pre-dose through 8 hours post-dose at Days 1 and 8
Population: PK Analysis Population includes all participants who are randomized, receive at least 1 study drug dose, and have PK samples collected for that period. Participants needed to have plasma concentration results at 3 or more time points beyond tmax (time to maximum measured plasma concentration) in order to have an evaluable estimate for λz
Measure: Mean (Standard Deviation); unit: 1/min
Arm/Group | Sublingual | Intramuscular
Number analyzed (Participants) | 41 | 46
1/min | 0.0042 (0.00077) | 0.0041 (0.00082)

13. Secondary Outcome: The Relative Bioavailability of Atropine Sulfate Administered SL Versus IM as Measured by Volume of Distribution (Vd/F)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 5, 10, 15, 20, 30, 45, 60, and 90 minutes, and 2, 2.5, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using noncompartmental analysis (NCA) methods.
  Vd/F is summarized by route of administration as the mean and standard deviation for all evaluable participants and expressed as mL.
Time Frame: Pre-dose through 8 hours post-dose at Days 1 and 8
Population: PK Analysis Population includes all participants who are randomized, receive at least 1 study drug dose, and have PK samples collected for that period. Participants needed to have plasma concentration results at 3 or more time points beyond tmax (time to maximum measured plasma concentration) in order to have an evaluable estimate for Vd/F.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Sublingual | Intramuscular
Number analyzed (Participants) | 41 | 46
mL | 447.17 (119.864) | 316.62 (88.157)

14. Secondary Outcome: The Relative Bioavailability of Atropine Sulfate Administered SL Versus IM as Measured by Total Body Clearance (CL/F)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 5, 10, 15, 20, 30, 45, 60, and 90 minutes, and 2, 2.5, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using noncompartmental analysis (NCA) methods.
  CL/F is summarized by route of administration as the mean and standard deviation for all evaluable participants and expressed as mL/min.
Time Frame: Pre-dose through 8 hours post-dose at Days 1 and 8
Population: PK Analysis Population includes all participants who are randomized, receive at least 1 study drug dose, and have PK samples collected for that period. Participants needed to have plasma concentration results at 3 or more time points beyond tmax (time to maximum measured plasma concentration) in order to have an evaluable estimate for CL/F.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Sublingual | Intramuscular
Number analyzed (Participants) | 41 | 46
mL/min | 1823.440 (420.5016) | 1248.156 (226.2500)

15. Secondary Outcome: The Relative Bioavailability of Atropine Sulfate Administered SL Versus IM as Measured by Absorption Rate Constant (Ka)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 5, 10, 15, 20, 30, 45, 60, and 90 minutes, and 2, 2.5, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using noncompartmental analysis (NCA) methods.
  Ka is summarized by route of administration as the mean and standard deviation for all evaluable participants and expressed 1/min.
Time Frame: Pre-dose through 8 hours post-dose at Days 1 and 8
Population: PK Analysis Population includes all participants who are randomized, receive at least 1 study drug dose, and have PK samples collected for that period. Participants needed to have plasma concentration results at 3 or more time points from pre-dose through tmax (time to maximum measured plasma concentration) in order to have an evaluable estimate for Ka
Measure: Mean (Standard Deviation); unit: 1/min
Arm/Group | Sublingual | Intramuscular
Number analyzed (Participants) | 45 | 44
1/min | 0.022 (0.0147) | 0.117 (0.2034)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were reported from the time the participant received the first dose of atropine at Day 1 until completion of the follow-up period at Day 15..
Description: Adverse events grade 1 or higher were recorded on the appropriate AE electronic case report form (eCRF) for this study. The study site graded the severity of AEs experienced by the study participants according to the criteria set forth in the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0.
Arm/Group | Sublingual | Intramuscular
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/46
Other Adverse Events (participants affected / at risk) | 14/45 | 22/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sublingual (N=45) | Intramuscular (N=46)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 12 (12) | 22 (22)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT06366087/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT06366087/SAP_001.pdf
  • Informed Consent Form (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT06366087/ICF_002.pdf